CLINICAL TRIAL: NCT06595199
Title: PRAMS: Peer-support To Reduce Antenatal Maternal Smoking: Development And Feasibility Testing Of A Social Media Group To Provide Peer Support And Enhance Quit Rates For Women Who Smoke In Pregnancy
Brief Title: PRAMS: Peer-support To Reduce Antenatal Maternal Smoking
Acronym: PRAMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University of Huddersfield (Other); National Institute for Health Research, United Kingdom (Other Government); The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1670751
Record Dates: First submitted 2024-08-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Smoking Cessation; Pregnancy Related
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: online group (Experimental): Online peer support group
  Interventions: Other: Online peer support
- Control: standard care (No Intervention): Standard care

INTERVENTIONS:
Other: Online peer support — A closed online peer support group
  Arms: Intervention: online group

SUMMARY:
The goal of this feasibility is test the feasibility of conducting a randomised trial of the use of an online peer support group to promote smoking cessation and enhance sustained abstinence for women who smoke in pregnancy.

Researchers will compare the group who receive the intervention (along side standard care) with a group who receive standard care alone.

DETAILED DESCRIPTION:
Participants will be asked to complete 2 questionnaires (and the intervention group will be asked to sign up to an online support group). They will be offered the opportunity to also take part in a follow up interview to explore acceptability and feasibility of the a future trial

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Smoking at beginning of pregnancy
* Access to mobile phone

Exclusion Criteria:

* Under 16 years of age

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 12 months
  Number of participants as % of smokers booked at the Trust
Attrition rate | 12 months
  How many participants complete all elements of the study

SECONDARY OUTCOMES:
Smoking status at end of pregnancy | 12 months
  Smoking status at end of pregnancy assessed by self report and cotinine testing
Engagement with stop smoking services | 12 months
  Record of initial and subsequent visits

IPD SHARING:
Plan to Share IPD: No
This is a feasibility study , so IPD not relevant